CLINICAL TRIAL: NCT00538005
Title: A Phase I/II Trial of Nexavar, Avastin and Eloxatin in Patients With Metastatic Malignant Melanoma
Brief Title: Sorafenib, Bevacizumab, and Oxaliplatin in Treating Patients With Metastatic Malignant Melanoma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: San Diego Pacific Oncology & Hematology Associates (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000551557; POHA-0603
Record Dates: First submitted 2007-10-01; First posted 2007-10-02 (Estimated); Last update posted 2014-01-10 (Estimated); Status verified 2009-07

CONDITIONS: Melanoma (Skin)
Keywords: recurrent melanoma; stage IV melanoma
MeSH Terms: conditions — Melanoma | interventions — Bevacizumab; Oxaliplatin; Sorafenib

INTERVENTIONS:
Biological: bevacizumab
Drug: oxaliplatin
Drug: sorafenib tosylate

SUMMARY:
RATIONALE: Sorafenib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Bevacizumab may also stop the growth of malignant melanoma by blocking blood flow to the tumor. Drugs used in chemotherapy, such as oxaliplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving sorafenib together with bevacizumab and oxaliplatin may kill more tumor cells.

PURPOSE: This phase I/II trial is studying the side-effects and best dose of sorafenib when given together with bevacizumab and oxaliplatin and to see how well it works in treating patients with metastatic malignant melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine the maximum tolerated dose of sorafenib tosylate when administered with bevacizumab and oxaliplatin.
* To determine the effect of this treatment regimen on the complete and partial response rate in patients with metastatic melanoma.
* To determine the effect of this treatment regimen on the progression-free and overall survival of patients with metastatic melanoma.

OUTLINE: This is a phase I dose-escalation study of sorafenib tosylate followed by a phase II study.

* Phase I: Patients receive bevacizumab IV over 30-90 minutes and oxaliplatin IV over 2 hours on day 1. Patients also receive oral sorafenib tosylate twice daily on days 1-14. Treatment repeats every 2 weeks in the absence of disease progression or unacceptable toxicity.
* Phase II: Patients receive sorafenib tosylate at the maximum tolerated dose and bevacizumab and oxaliplatin as in phase I.

After completion of study therapy, patients are followed for at least 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed melanoma

  * Metastatic disease
* Measurable or evaluable non-CNS disease

  * Measurable disease, defined as a unidimensionally measurable lesion as determined by physical exam, x-ray, CT scan, MRI, or other radiographic procedure
  * Evaluable disease, defined as a lesion that can be seen radiographically but is not unidimensionally measurable

    * Previously irradiated lesions with documented progression are allowed provided there are no other sites of metastatic disease
* No active brain metastases

  * Previously treated, responding brain metastases allowed, provided there is measurable disease outside of the CNS

    * At least 3 weeks since prior chemotherapy and 6 weeks since prior radiotherapy for CNS disease

PATIENT CHARACTERISTICS:

Inclusion criteria:

* ECOG performance status 0-2
* Life expectancy ≥ 3 months
* ANC ≥ 1,200/mm^3
* Platelet count ≥ 100,000/mm^3
* Creatinine ≤ 1.5 mg/dL OR creatinine clearance ≥ 50 mL/min
* Bilirubin ≤ 3.0 mg/dL
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* EKG with no evidence of serious arrhythmia or recent myocardial infarction

Exclusion criteria:

* Active infection
* Chronic underlying immunodeficiency disease
* Other serious concurrent illness
* Other forms of cancer within 5 years of initial diagnosis except nonmelanoma skin cancer and cervical cancer
* Congestive heart failure or myocardial infarction within the past 6 months

PRIOR CONCURRENT THERAPY:

Inclusion criteria:

* See Disease Characteristics
* At least 6 weeks since prior radiotherapy
* More than 4 weeks since prior surgery
* Prior biologic therapy allowed

Exclusion criteria:

* Prior cytotoxic agents
* Prior sorafenib tosylate, bevacizumab, or oxaliplatin
* Concurrent biological therapy, except growth factors for anemia, neutropenia, or thrombocytopenia
* Concurrent radiotherapy, chemotherapy, or surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2007-05; Primary Completion 2009-07 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose of sorafenib tosylate when administered with bevacizumab and oxaliplatin
Response (complete and partial) as assessed by RECIST criteria
Progression-free survival
Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Edward F. McClay, MD, Principal Investigator — San Diego Pacific Oncology & Hematology Associates
Locations (1):
- San Diego Pacific Oncology and Hematology Associates, Incorporated - Encinitas, Encinitas, California, United States